CLINICAL TRIAL: NCT05925062
Title: Effect of a Mental Wellness App on the Mental Wellness of Medical and Nurse Anesthesia Students
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study team concluded that it was unlikely that the study population would be adherent to the tool planned for the study and therefore the study would not be valuable to pursue.
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00098397
Record Dates: First submitted 2023-06-20; First posted 2023-06-29 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Mental Health Issue
Keywords: stress levels; anxiety; depression
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: This will be a non-randomized, control-group, year-long study exploring the impact of a mental wellness app on various aspects of mental wellness in first-year medical students and second-year nurse anesthesia (CRNA) students from Wake Forest University School of Medicine (WFUSM) during the 2023 - 2024 academic year (approximately July 2023 - June 2024).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QActual (Experimental): QActual is a phone-based app that offers peer-to-peer support, tracks mental wellness self-assessments, and provides support to users who are in crisis.
  Interventions: Behavioral: QActual
- Control Arm - Subjects not using App (No Intervention): No intervention

INTERVENTIONS:
Behavioral: QActual — QActual is a phone-based app that offers peer-to-peer support, tracks mental wellness self-assessments, and provides support to users who are in crisis.
  Arms: QActual

SUMMARY:
Mental health issues and suicide are becoming increasingly common among health care trainees and providers. Suicide is the leading cause of death among male medical residents and the second leading cause of death among female residents.

DETAILED DESCRIPTION:
Training programs are usually very rigorous, caring for patients is stressful, and those who care for others often feel that they can't or shouldn't admit that they need care themselves. Unfortunately, there is often a stigma associated with mental illness, and trainees may feel that admitting that they struggle could damage their careers. The need exists for easily accessible, immediate, crisis support for medical trainees who are experiencing a mental health crisis. Although the effectiveness of mental health apps has been evaluated in college students, there is very little data assessing their use in medical and nurse anesthesia students. The purpose of this study is to evaluate the effect of a mental wellness app on the mental wellness of medical and nurse anesthesia students.

ELIGIBILITY:
Inclusion Criteria:

* first-year medical students and second-year nurse anesthesia (CRNA) students from Wake Forest University School of Medicine during the 2023 - 2024 academic year (approximately July 2023 - June 2024).

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-07 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire-9 (PHQ-9) scores | Baseline
  Scores less than 5 almost always signified the absence of a depressive disorder; scores of 5 to 9 predominantly represented patients with either no depression or subthreshold (i.e., other) depression; scores of 10 to 14 represented a spectrum of patients; and scores of 15 or greater usually indicated major depression.
Patient Health Questionnaire-9 (PHQ-9) scores | Month 3
  Scores less than 5 almost always signified the absence of a depressive disorder; scores of 5 to 9 predominantly represented patients with either no depression or subthreshold (i.e., other) depression; scores of 10 to 14 represented a spectrum of patients; and scores of 15 or greater usually indicated major depression.
Patient Health Questionnaire-9 (PHQ-9) scores | Month 6
  Scores less than 5 almost always signified the absence of a depressive disorder; scores of 5 to 9 predominantly represented patients with either no depression or subthreshold (i.e., other) depression; scores of 10 to 14 represented a spectrum of patients; and scores of 15 or greater usually indicated major depression.
Patient Health Questionnaire-9 (PHQ-9) scores | Month 9
  Scores less than 5 almost always signified the absence of a depressive disorder; scores of 5 to 9 predominantly represented patients with either no depression or subthreshold (i.e., other) depression; scores of 10 to 14 represented a spectrum of patients; and scores of 15 or greater usually indicated major depression.
Patient Health Questionnaire-9 (PHQ-9) scores | Year 1
  Scores less than 5 almost always signified the absence of a depressive disorder; scores of 5 to 9 predominantly represented patients with either no depression or subthreshold (i.e., other) depression; scores of 10 to 14 represented a spectrum of patients; and scores of 15 or greater usually indicated major depression.

SECONDARY OUTCOMES:
Number of crisis alerts triggered | Year 1
  Number of crisis alerts triggered
Number of daily wellness check-ins completed | Year 1
  Number of daily wellness check-ins completed
Satisfaction with the app Scores | Year 1
  Satisfaction with the app scores - a global scale that is used to assess attitudes and views. It is a scale with 5 answer options which has two utmost poles and a neutral option linked with intermediate answer options. For example, agree, fully agree, neither agree nor disagree, disagree, and fully disagree
Time periods associated with lower daily wellness check scores | Year 1
  Time periods associated with lower daily wellness check scores (these will be compared to the academic calendar to detect any correlations) - The mean daily wellness check scores for Medical students and CRNA students will be retrospectively reviewed. Days where the mean score for the day differ significantly from the mean score for the year will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: James R Beardsley, PharmD, BCPS, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No